CLINICAL TRIAL: NCT06254157
Title: Generalized Anxiety Disorder Clinical Trials: An Analysis Regarding Engagement Trends and Participation of Generalized Anxiety Disorder Patients Involved in Clinical Trials
Brief Title: Understanding of Participation Trends Within Generalized Anxiety Disorder Patients Involved in Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 57777066
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: generalized anxiety disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Typically, certain demographic groups tend to participate more in medical research. However, there is insufficient research explaining the trial characteristics that influence the involvement of these specific demographics.

This study aims to collect extensive data on the clinical trial experiences of individuals with generalized anxiety disorder. The goal is to identify the factors that hinder a patient's enrollment or completion of a trial.

Additionally, the research will examine the data from various demographic perspectives to identify recurring patterns that could offer valuable insights for future generalized anxiety disorder patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of generalized anxiety disorder
* Participant must be 18 years of age or older
* Participant must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study.

Exclusion Criteria:

* Pregnant or lactating woman
* Participant is actively receiving study therapy in another
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with generalized anxiety disorder who are actively contemplating involvement in a clinical trial but have not yet completed the enrollment and randomization process.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a generalized anxiety disorder clinical research. | 3 months
Number of generalized anxiety disorder study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slee A, Nazareth I, Bondaronek P, Liu Y, Cheng Z, Freemantle N. Pharmacological treatments for generalised anxiety disorder: a systematic review and network meta-analysis. Lancet. 2019 Feb 23;393(10173):768-777. doi: 10.1016/S0140-6736(18)31793-8. Epub 2019 Jan 31. PMID 30712879
- [Background] Hofmann SG, Smits JA. Cognitive-behavioral therapy for adult anxiety disorders: a meta-analysis of randomized placebo-controlled trials. J Clin Psychiatry. 2008 Apr;69(4):621-32. doi: 10.4088/jcp.v69n0415. PMID 18363421
- [Background] Santiago J, Akeman E, Kirlic N, Clausen AN, Cosgrove KT, McDermott TJ, Mathis B, Paulus M, Craske MG, Abelson J, Martell C, Wolitzky-Taylor K, Bodurka J, Thompson WK, Aupperle RL. Protocol for a randomized controlled trial examining multilevel prediction of response to behavioral activation and exposure-based therapy for generalized anxiety disorder. Trials. 2020 Jan 6;21(1):17. doi: 10.1186/s13063-019-3802-9. PMID 31907032

DOCUMENTS (1):
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT06254157/ICF_000.pdf